CLINICAL TRIAL: NCT00905281
Title: Randomized Controlled Trial Assessing the Impact of Routine "Oncologist-supportive Care Team" Consultation on the Use of an Additional Line of Chemotherapy in Metastatic Breast Cancer Patients
Brief Title: Study of Impact of Routine "Clinical Cancer Department/Supportive Care Department" Consultation on the Prescription of an Additional Line of Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSS; ET 2007-037
Record Dates: First submitted 2009-05-05; First posted 2009-05-20 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Supportive care; Third or fourth line of chemotherapy; Quality of life; Treatment preferences
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Action Group (Experimental)
  Interventions: Other: Action Group
- Standard care (Other)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Action Group — On inclusion, a visit will be organized between the patient and at least 2 members of the DISSPO staff. It will allow an evaluation of supportive care needs and the proposition of a personalized care plan.
  Then, a consultation between the referring oncologist and the DISSPO will be organized once a month, so that the personalized care plan could be adapted if necessary.
  Arms: Action Group
Other: Standard care — No specific intervention
  Arms: Standard care

SUMMARY:
The purpose of this study is to assess the impact of systematic "clinical cancer department/supportive care department" consultation meetings, versus standard care, on the prescription of an additional line of chemotherapy in patients with metastatic breast cancer and visceral involvement after 3 or 4 lines of chemotherapy.

This is a prospective paucicentric open label randomized controlled study with 2 parallel arms.

Eligible patients will be randomly assigned to either arm "Study group" or "Standard care".

The number of patients required to demonstrate a 30% reduction of the number of prescriptions for an additional line chemotherapy, assuming an alpha risk of 5% and 80% power, is 100 (50 in each arm).

DETAILED DESCRIPTION:
The hypothesis tested is that systematic routine consultation between the supportive care team and clinical oncologists will allow more efficient utilization of supportive care by metastatic breast cancer patients, and will reduce the isolation of physicians involved in the management of these patients. Physicians will then be able to help the patients make realistic decisions for the best possible quality of life and in full accordance with their preferences.

The DISSPO (Department of Interdisciplinary Supportive Care for Cancer Patients) focuses on psycho-oncology, pain evaluation and treatment, palliative care, social service, dietary guidance and physiotherapy. Usually, visits with the DISSPO are arranged when the patients need supportive care but are not included in routine care. In this study, contacts between clinical oncologists and supportive care staff will be formalized and systematized. A specific visit called "supportive care visit" will be organized to investigate the needs of the patient so that a personalized care plan can be proposed. Moreover, a consultation between the referring oncologist and the DISSPO will be organized at least once a month.

Besides the main objective of this study (see brief summary), there are secondary objectives which are to evaluate the impact of systematic "Clinical cancer department/Supportive care department" consultation meetings versus standard care on:

* the use of supportive care
* symptom control
* anxiety-depression levels
* quality of life
* patient representations (adaptation to the disease and locus of control)
* patient perception of social support
* patient satisfaction with the care
* impact of disease on the family
* satisfaction of the referring oncologist

ELIGIBILITY:
Inclusion Criteria:

* Woman aged >= 18 years
* Metastatic breast cancer with visceral involvement
* Patient requiring a 3rd or a 4th line of chemotherapy
* Patient followed at Léon Bérard Cancer Center
* Patient affiliated with social security
* Patient able to read and write French
* Written, voluntary, informed consent

Exclusion Criteria:

* Ongoing chemotherapy other than third or fourth line
* Only skin or bone metastasis
* Follow-up impossible for social, geographical, familial or psychological reasons
* Patient deprived of freedom
* Pregnant or lactating woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Rate of prescriptions for a 4th or 5th line of chemotherapy | At the time of progression on 3rd or 4th line of chemotherapy.
  When patients progress under 3rd or 4th line of chemotherapy, rate of prescriptions for a 4th or 5th line will be collected.

SECONDARY OUTCOMES:
Evaluation of the number and type of DISSPO interventions | During the period of inclusion in the study: between the inclusion and the time of progression on 3rd or 4th line of chemotherapy
Self-evaluation of symptom control using the Edmonton scale | Self-administered questionnaire at inclusion, at 6 months and 12 months post-inclusion, at the end and 3 months after the end of the 3rd or 4th line of chemotherapy
Self-rating of anxiety-depression using the HADS scale | Self-administered questionnaire at inclusion, at 6 months and 12 months post-inclusion, at the end and 3 months after the end of the 3rd or 4th line of chemotherapy.
Self-evaluation of quality of life using the QLQC30 scale. | Self-administered questionnaire at inclusion, at 6 months and 12 months post-inclusion, at the end and 3 months after the end of the 3rd or 4th line of chemotherapy.
Self-evaluation of adaptation and of the locus of control using the CLCS scale. | Self-administered questionnaire at inclusion, at 6 months and 12 months post-inclusion, at the end and 3 months after the end of the 3rd or 4th line of chemotherapy.
Self-evaluation of social support using the QSSP scale | Self-administered questionnaire at inclusion, at 6 months and 12 months post-inclusion, at the end and 3 months after the end of the 3rd or 4th line of chemotherapy.
Self-evaluation of satisfaction with care using the F-PMH/PSQ MD scale | Self-administered questionnaire at inclusion, at 6 months and 12 months post-inclusion, at the end and 3 months after the end of the 3rd or 4th line of chemotherapy.
Self-evaluation of the impact of disease on family using the GHQ28 scale | Self-administered questionnaire at inclusion, at 6 months and 12 months post-inclusion, at the end and 3 months after the end of the 3rd or 4th line of chemotherapy.
Self-evaluation of satisfaction by the referring physician using the Likert scale | Self-administered questionnaire at 6 months and 12 months post-inclusion, at the end and 3 months after the end of the 3rd or 4th line of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: CHVETZOFF Gisèle, MD, Principal Investigator — Centre Leon Berard
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

REFERENCES:
- [Background] Gennari A, Conte P, Rosso R, Orlandini C, Bruzzi P. Survival of metastatic breast carcinoma patients over a 20-year period: a retrospective analysis based on individual patient data from six consecutive studies. Cancer. 2005 Oct 15;104(8):1742-50. doi: 10.1002/cncr.21359. PMID 16149088
- [Background] Slamon DJ, Leyland-Jones B, Shak S, Fuchs H, Paton V, Bajamonde A, Fleming T, Eiermann W, Wolter J, Pegram M, Baselga J, Norton L. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001 Mar 15;344(11):783-92. doi: 10.1056/NEJM200103153441101. PMID 11248153
- [Background] Giordano SH, Buzdar AU, Smith TL, Kau SW, Yang Y, Hortobagyi GN. Is breast cancer survival improving? Cancer. 2004 Jan 1;100(1):44-52. doi: 10.1002/cncr.11859. PMID 14692023
- [Background] Banerji U, Kuciejewska A, Ashley S, Walsh G, O'Brien M, Johnston S, Smith I. Factors determining outcome after third line chemotherapy for metastatic breast cancer. Breast. 2007 Aug;16(4):359-66. doi: 10.1016/j.breast.2007.01.004. Epub 2007 May 16. PMID 17509879
- [Background] Rha SY, Moon YH, Jeung HC, Kim YT, Sohn JH, Yang WI, Suh CO, Kim GE, Roh JK, Chung HC. Gemcitabine monotherapy as salvage chemotherapy in heavily pretreated metastatic breast cancer. Breast Cancer Res Treat. 2005 Apr;90(3):215-21. doi: 10.1007/s10549-004-2468-4. PMID 15830134
- [Background] Dufresne A, Pivot X, Tournigand C, Facchini T, Altweegg T, Chaigneau L, De Gramont A. Impact of chemotherapy beyond the first line in patients with metastatic breast cancer. Breast Cancer Res Treat. 2008 Jan;107(2):275-9. doi: 10.1007/s10549-007-9550-7. Epub 2007 Mar 23. PMID 17380382
- [Background] Detmar SB, Muller MJ, Schornagel JH, Wever LD, Aaronson NK. Role of health-related quality of life in palliative chemotherapy treatment decisions. J Clin Oncol. 2002 Feb 15;20(4):1056-62. doi: 10.1200/JCO.2002.20.4.1056. PMID 11844830
- [Background] Weeks JC, Cook EF, O'Day SJ, Peterson LM, Wenger N, Reding D, Harrell FE, Kussin P, Dawson NV, Connors AF Jr, Lynn J, Phillips RS. Relationship between cancer patients' predictions of prognosis and their treatment preferences. JAMA. 1998 Jun 3;279(21):1709-14. doi: 10.1001/jama.279.21.1709. PMID 9624023
- [Background] Slevin ML, Stubbs L, Plant HJ, Wilson P, Gregory WM, Armes PJ, Downer SM. Attitudes to chemotherapy: comparing views of patients with cancer with those of doctors, nurses, and general public. BMJ. 1990 Jun 2;300(6737):1458-60. doi: 10.1136/bmj.300.6737.1458. PMID 2379006
- [Background] Glare P, Virik K, Jones M, Hudson M, Eychmuller S, Simes J, Christakis N. A systematic review of physicians' survival predictions in terminally ill cancer patients. BMJ. 2003 Jul 26;327(7408):195-8. doi: 10.1136/bmj.327.7408.195. PMID 12881260
- [Background] Asola R, Huhtala H, Holli K. Intensity of diagnostic and treatment activities during the end of life of patients with advanced breast cancer. Breast Cancer Res Treat. 2006 Nov;100(1):77-82. doi: 10.1007/s10549-006-9224-x. Epub 2006 Jun 7. PMID 16758120
- [Background] Braga S, Miranda A, Fonseca R, Passos-Coelho JL, Fernandes A, Costa JD, Moreira A. The aggressiveness of cancer care in the last three months of life: a retrospective single centre analysis. Psychooncology. 2007 Sep;16(9):863-8. doi: 10.1002/pon.1140. PMID 17245696
- [Background] A controlled trial to improve care for seriously ill hospitalized patients. The study to understand prognoses and preferences for outcomes and risks of treatments (SUPPORT). The SUPPORT Principal Investigators. JAMA. 1995 Nov 22-29;274(20):1591-8. PMID 7474243
- [Background] Chvetzoff G, Perol D, Devaux Y, Lancry L, Rebattu P, Magnet M, Dubost E, Bertrand M, Garcon C, Thevenet G, Gobet S, Arbiol E, Saltel P. [Prospective study on the quality of care and quality of life in advanced cancer patients treated at home or in hospital: intermediate analysis of the Trapado study]. Bull Cancer. 2006 Feb;93(2):213-21. French. PMID 16517418
- [Background] Homsi J, Walsh D, Nelson KA, LeGrand SB, Davis M, Khawam E, Nouneh C. The impact of a palliative medicine consultation service in medical oncology. Support Care Cancer. 2002 May;10(4):337-42. doi: 10.1007/s00520-002-0341-8. Epub 2002 Feb 15. PMID 12029434
- [Background] Manfredi PL, Morrison RS, Morris J, Goldhirsch SL, Carter JM, Meier DE. Palliative care consultations: how do they impact the care of hospitalized patients? J Pain Symptom Manage. 2000 Sep;20(3):166-73. doi: 10.1016/s0885-3924(00)00163-9. PMID 11018334
- [Background] McLachlan SA, Allenby A, Matthews J, Wirth A, Kissane D, Bishop M, Beresford J, Zalcberg J. Randomized trial of coordinated psychosocial interventions based on patient self-assessments versus standard care to improve the psychosocial functioning of patients with cancer. J Clin Oncol. 2001 Nov 1;19(21):4117-25. doi: 10.1200/JCO.2001.19.21.4117. PMID 11689579
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Cousson-Gelie F, Irachabal S, Bruchon-Schweitzer M, Dilhuydy JM, Lakdja F. Dimensions of cancer locus of control scale as predictors of psychological adjustment and survival in breast cancer patients. Psychol Rep. 2005 Dec;97(3):699-711. doi: 10.2466/pr0.97.3.699-711. PMID 16512284
- [Background] Bolognini M, Bettschart W, Zehnder-Gubler M, Rossier L. The validity of the French version of the GHQ-28 and PSYDIS in a community sample of 20 year olds in Switzerland. Eur Arch Psychiatry Neurol Sci. 1989;238(3):161-8. doi: 10.1007/BF00451005. PMID 2721534
- [Background] Barlesi F, Chabert-Greillier L, Loundou A, Simeoni MC, Greillier L, Doddoli C, Astoul P, Auquier P. [Validation of the French version of the Princess Margaret Hospital Patient Satisfaction with their Doctor Questionnaire]. Rev Mal Respir. 2006 Jun;23(3 Pt 1):227-36. doi: 10.1016/s0761-8425(06)71572-8. French. PMID 16788523
- [Background] O'Mahony S, Blank AE, Zallman L, Selwyn PA. The benefits of a hospital-based inpatient palliative care consultation service: preliminary outcome data. J Palliat Med. 2005 Oct;8(5):1033-9. doi: 10.1089/jpm.2005.8.1033. PMID 16238516
- [Background] Virik K, Glare P. Profile and evaluation of a palliative medicine consultation service within a tertiary teaching hospital in Sydney, Australia. J Pain Symptom Manage. 2002 Jan;23(1):17-25. doi: 10.1016/s0885-3924(01)00371-2. PMID 11779664
- [Background] Fleiss JL, Tytun A, Ury HK. A simple approximation for calculating sample sizes for comparing independent proportions. Biometrics. 1980 Jun;36(2):343-6. PMID 26625475
- [Background] Schemper M, Smith TL. A note on quantifying follow-up in studies of failure time. Control Clin Trials. 1996 Aug;17(4):343-6. doi: 10.1016/0197-2456(96)00075-x. No abstract available. PMID 8889347
- [Background] Kleinbaum DG, Klein M. In: Springer N-Y. Logistic regression. A Self-Learning Text. 2002
- [Background] In: EORTC Quality of Life Study Group. Brussels. EORTC QLQC-30 scoring manual, 2nd ed. 1999
- [Background] Osoba D, Bezjak A, Brundage M, Zee B, Tu D, Pater J; Quality of Life Committee of the NCIC CTG. Analysis and interpretation of health-related quality-of-life data from clinical trials: basic approach of The National Cancer Institute of Canada Clinical Trials Group. Eur J Cancer. 2005 Jan;41(2):280-7. doi: 10.1016/j.ejca.2004.10.017. PMID 15661554
- [Derived] Chvetzoff G, Bouleuc C, Lardy-Cleaud A, Saltel P, Dieras V, Morelle M, Guastalla JP, Tredan O, Rebattu P, Pop S, Ray-Coquard I, Pierga JY, Mignot L, Laurence V, Bourne-Branchu V, Perol D, Bachelot T. Impact of early palliative care on additional line of chemotherapy in metastatic breast cancer patients: results from the randomized study OSS. Support Care Cancer. 2022 Dec 27;31(1):82. doi: 10.1007/s00520-022-07561-x. PMID 36574052